CLINICAL TRIAL: NCT05972551
Title: A Phase 3, Open-Label, Multicenter, Randomized Study to Evaluate Efficacy and Safety of Romosozumab Compared With Bisphosphonates in Children and Adolescents With Osteogenesis Imperfecta
Brief Title: Study to Evaluate Efficacy and Safety of Romosozumab Compared With Bisphosphonates in Children and Adolescents With Osteogenesis Imperfecta
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200105; 2023-503294-37 (EudraCT Number)
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Romosozumab; EVENITY®; Bisphosphonates
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — romosozumab; Diphosphonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romosozumab (Experimental): Participants will receive romosozumab once a month (QM) for 12 months.
  Interventions: Drug: Romosozumab
- Standard of Care Bisphosphonate (Active Comparator): Participants will receive bisphosphonates per local standard of care treatment regimens, as determined by the investigator for 12 months.
  Interventions: Drug: Bisphosphonate

INTERVENTIONS:
Drug: Romosozumab — Subcutaneous (SC) injection
  Other Names: EVENITY®
  Arms: Romosozumab
Drug: Bisphosphonate — Administration determined by investigator according to the local standard of care
  Arms: Standard of Care Bisphosphonate

SUMMARY:
The primary objective of this study is to evaluate the effect of romosozumab treatment for 12-months compared with bisphosphonate(s) on the number of clinical fractures at 12-months; the number of any fractures at 12-months and change in lumbar spine bone mineral density (BMD) Z-score at 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study specific activities/procedures.

OR

* Participant's legally authorized representative has provided informed consent when the participant is legally too young to provide informed consent and the participant has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated.
* Ambulatory male and female children and adolescents, age 5 to <18 years, including ambulatory with assistance as defined in the pediatric osteogenesis imperfecta (OI) population.
* Clinical diagnosis of OI, defined as clinical history consistent with type I, III, or IV OI as determined by presence of expected phenotype (examples include: facial shape, voice, blue sclera, dentinogenesis imperfecta, typical radiographic features, fracture pattern) and lack of additional features unrelated to type I, III, or IV OI (eg, blindness, mental retardation, neuropathy, and craniosynostosis).

  o If familial, also must be autosomal dominant.
* Meets at least one of the following:

  * 3 or more fractures within the previous 2 years, or
  * 1 or more nonvertebral fracture(s) within the previous 2 years and at least 1 prevalent vertebral fracture, or
  * 2 or more prevalent vertebral fractures.

Exclusion Criteria:

Disease Related

* History of an electrophoresis pattern inconsistent with type I, III or IV OI.
* History of known mutation in a gene other than collagen type I alpha 1/collagen type I alpha 2 (COL1A1/COL1A2) causing OI or other metabolic bone disease.
* History of congenital dislocation of the radial head, interosseous membrane calcification, or exuberant callus formation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Number of Clinical Fractures | 12 months
  Clinical fractures include clinical vertebral fractures and nonvertebral fractures.
Number of Any Fractures | 12 months
  Fractures include new and worsening vertebral compression fractures, whether clinically silent or manifest, and nonvertebral fractures.
Change from Baseline in Lumbar Spine BMD Z-score at 12 Months, as assessed by DXA | Baseline and 12 months

SECONDARY OUTCOMES:
Change from Baseline in lumbar spine BMD Z-score at 6 months and 12 months, as assessed by DXA | Baseline, 6 months, and 12 months
Change from Baseline in Total Hip BMD Z-score at 6 Months and at 12 Months, as assessed by DXA | Baseline, 6 months, and 12 months
Change from Baseline in Femoral Neck BMD Z-score at 6 Months and at 12 Months, as assessed by DXA | Baseline, 6 months, and 12 months
Number of Participants with Any Fractures | 12 months
Number of Participants with Clinical Fractures | 12 months
Number of Participants with New or Worsening Vertebral Fractures | 12 months
Number of Participants with Nonvertebral Fractures | 12 months
Number of Participants with Long Bone Fractures | 12 months
Number of New or Worsening Vertebral Fractures | 12 months
Number of Nonvertebral Fractures | 12 months
Number of Long Bone Fractures | 12 months
Change from Baseline in Child Health Questionnaire - Parent Version (CHQ-PF-50) Physical Summary Score | Baseline and 12 months
  The CHQ-PF-50 measures how a child's condition affects their ability to function in daily life. The CHQ-PF-50 measures 50 items in the following domains: physical functioning, role/social limitations - physical, general health perceptions, bodily pain/discomfort, family activities, role/social limitations - emotional/behavioral, parent impact - time, parent impact - emotion, self-esteem, mental health, behavior, family cohesion, change in health.
  Each item is rated on a scale from "without any difficulty" to "unable to do". Total scores for each item are transformed to 0 - 100 scale, with lower scores indicating worse health states. Higher change from baseline scores indicate better or more positive health states.
Change from Baseline in Childhood Health Assessment Questionnaire (CHAQ) Disability Score | Baseline and 12 months
  The CHAQ measures how a child's condition affects their ability to function in daily life. The CHAQ measures 50 items in the following domains: physical functioning, role/social limitations - physical, general health perceptions, bodily pain/discomfort, family activities, role/social limitations emotional/behavioral, self-esteem, mental health, behavior, family cohesion, change in health.
  Each item is rated on a scale from "without any difficulty" to "unable to do". Total scores for each item are transformed to 0 - 100 scale, with lower scores indicating worse health states. Higher change from baseline scores indicate better or more positive health states.
Change from Baseline in the Wong-Baker Faces Pain Rating Scale | Baseline and 12 months
  The Wong-Baker Faces Pain Rating Scale is a horizontal pain scale that consists of six hand-drawn faces that range from a smiling "no hurt" face with a score of 0 to a crying "hurts worst" face with a score of 10. Greater change from baseline scores indicate greater pain experienced by the participant.
Serum Concentration of Romosozumab | Day 1 to Month 12
Number of Participants who Experience Treatment-emergent Adverse Events (TEAEs) at 12 Months | 12 months
  Any clinically signification change from baseline in laboratory values and vital signs after first dose will be recorded as a TEAE.
Number of Participants who Experience TEAEs from Month 12 to Month 15 | Month 12 to Month 15
  Any clinically signification change from baseline in laboratory values and vital signs after first dose will be recorded as a TEAE.
Number of Participants with Anti-drug Antibodies (ADA) to Romosozumab | Up to 15 months
Number of Participants who Experience TEAEs at 15 Months | 15 months
  Any clinically signification change from baseline in laboratory values and vital signs after first dose will be recorded as a TEAE.
Number of Participants with a Narrowing from Baseline to 6 Months in the Intracranial Nerve Tract in the Cranium and Vault of the Skull | Baseline and 6 months
  Measured in a subset of participants who receive cranial nerve computerized tomography (CT) scans.
Number of Participants with a Narrowing from Baseline to 12 Months in the Intracranial Nerve Tract in the Cranium and Vault of the Skull | Baseline and 12 months
  Measured in a subset of participants who receive cranial nerve CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (60):
- United States (14):
  - Childrens Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of California, Los Angeles Interventional Clinical Trials, Los Angeles, California
  - Nemours Hospital for Children, Wilmington, Delaware
  - Nemours Childrens Hospital, Orlando, Florida
  - University of South Florida - Carol and Frank Morsani Center for Advanced Health Care, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - Mayo Clinic Childrens Center, Rochester, Minnesota
  - Gillette Childrens Hospital and Clinic Saint Paul, Saint Paul, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Marshfield Clinic, Marshfield, Wisconsin
- Australia (2):
  - Monash Childrens Hospital, Clayton, Victoria
  - Perth Childrens Hospital, Nedlands, Western Australia
- Kepler Universitaetsklinikum GmbH, Linz, Austria
- Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Belgium
- Canada (3):
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec
- China (8):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Tongji Hospital , Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Childrens Hospital of Soochow University, Suzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Shanghai Sixth Peoples Hospital, Shanghai
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Pellegrin, Bordeaux
  - Hopital Necker Enfants Malades, Paris
- Germany (2):
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Wuerzburg, Würzburg
- Semmelweis Egyetem, Budapest, Hungary
- Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona, Italy
- Japan (4):
  - Okayama Saiseikai Outpatient Center Hospital, Okayama, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka Womens and Childrens Hospital, Izumi-shi, Osaka
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
- Poland (5):
  - Centermed Krakow Sp zoo, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Centralny Szpital Kliniczny UMeds, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Centrum Medyczne Medyk Spolka z Ograniczona Odpowiedzialnoscia Spolka Komandytowa, Rzeszów
  - Szpital Miejski w Tychach Spolka z ograniczona odpowiedzialnoscia, Tychy
- Narodny ustav detskych chorob, Bratislava, Slovakia
- Spain (6):
  - Hospital de Cruces, Barakaldo, Basque Country
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Infantil Niño Jesus, Madrid
- Switzerland (2):
  - Universitaets-Kinderspital beider Basel, Basel
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Turkey (Türkiye) (4):
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Karadeniz Teknik Universitesi Tip Fakultesi, Trabzon
- United Kingdom (3):
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Manchester Childrens Hospital, Manchester
  - Sheffield Childrens Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com